CLINICAL TRIAL: NCT05482100
Title: CLinical Utility of the omnigrAf® biomarkeR Panel In The Care of kidneY Transplant Recipients
Acronym: CLARITY
Status: Not yet recruiting | Type: Observational
Sponsor: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TGRP11
Record Dates: First submitted 2022-07-18; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Kidney Transplant Rejection
Keywords: Biomarkers; Subclinical Rejection; Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients monitored with OmniGraf Testing: Subjects will have OmniGraf™ testing at study enrollment and thereafter every 3 months or at the same time as standard routine labs (minimum two per year). In addition, subjects will have OmniGraf™ testing at any time there is a workup for clinical events and referral to advanced care (transplant center, biopsy, etc)
  Interventions: Diagnostic Test: Patients monitored with OmniGraf testing

INTERVENTIONS:
Diagnostic Test: Patients monitored with OmniGraf testing — This is an observational study there are no protocol mandated interventions. OmniGraf results will be utilized in conjunction with standard of care assessments to determine patient management.

SUMMARY:
This is a prospective, multi-site, observational study with a matched control group. The primary objective is to evaluate change in renal function over time in recipients of kidney transplants who are undergoing OmniGrafTM monitoring in conjunction with patient medication-related burden monitoring.

DETAILED DESCRIPTION:
The survival benefits of solid organ transplants in the United States are well documented. Improvements in immunosuppression, better anti-microbial agents, and other aspects of ancillary care have resulted in significant improvements in short- term outcomes; however, there has been little improvement in long-term graft loss. A more recent analysis found that 65% of hospital readmissions in kidney transplant recipients had adverse drug events (ADE) considered contributory, and ADE-associated readmissions had a significantly higher hazard or graft loss and death compared to patients with readmissions not associated with an ADE. Even with knowledge of ADEs, clinicians may be reluctant to adjust immunosuppressive medications due to concerns of rejection risk during the period of medication adjustment. The OmniGrafTM biomarker panel (Transplant Genomics, Inc, Framingham, MA) includes the TruGraf® peripheral blood expression profile and the TRAC donor-derived cell-free DNA(dd-cfDNA) test, which have demonstrated a strong ability to identify immune quiescence in stable patients post kidney transplant, with a NPV of 94% when both tests are negative and a PPV of 89% for subclinical rejection when both tests are positive. Because of the strong "rule out" capabilities of OmniGrafTM, it would be an ideal complement to real-time ADE knowledge to help guide clinicians' decisions to adjust, or not adjust, the immunosuppressive regimen, and help provide a dialogue between patients and clinicians on the risk-benefit of medication adjustments. The aim of this study is to evaluate change in renal function over time in recipients of kidney transplants who are undergoing OmniGrafTM monitoring in conjunction with patient medication-related burden monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization;
* At least 18 years of age;
* Recipient of a primary or subsequent deceased-donor or living-donor kidney transplant;
* Between 3 months and 2 years post-transplant;
* Selected by provider to undergo OmniGraf™ testing as part of usual post-transplant care

Exclusion Criteria:

* Recipient of a combined organ transplant with an extra-renal organ and/or islet cell transplant;
* Recipient of a previous non-renal solid organ and/or islet cell transplant;
* Known to be pregnant;
* Known to be infected with Human Immunodeficiency Virus (HIV);
* Known to have active BK nephropathy;
* Known to have nephrotic proteinuria (per principal investigator); or
* Participation in other biomarker studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an observational study in adult (age ≥ 18 years), kidney transplant patients who are at 3 months to 2 years from the time of transplant. Approximately 500 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
GFR changes between study group and matched control group | 3 years
  Comparison of the slope change in estimated glomerular filtration rate (eGFR), calculated using the MDRD 4-variable equation and CKD-EPI, from baseline to the end of follow-up between study participants and a matched control group.

SECONDARY OUTCOMES:
PROMISE and Self efficacy results from baseline to study completion | 3 years
  Comparison of the Patient-Reported Outcomes Measurement Information System(PROMIS) Self-Efficacy for Managing Chronic Conditions - Managing Medications and Treatment-Short Form 4a (Self-Efficacy) at the end of follow-up to baseline PROMIS tools were developed to be disease non-specific measures of health-related domains. Each domain in composed of an item bank specific to a trait being measured. Item banks are calibrated on a common scale to facilitate comparability across varying populations. Depression is measured by various questions with answers ranging from never to always.
  Raw scores are transformed to standardized T-score metrics, with a mean of 50 and standard deviation of 10
PROMISE results from baseline to study completion | 3 years
  Comparison of the PROMIS-29 Profile v2.1 at the end of follow-up to baseline PROMIS tools were developed to be disease non-specific measures of health-related domains. Each domain in composed of an item bank specific to a trait being measured. Item banks are calibrated on a common scale to facilitate comparability across varying populations. Depression is measured by various questions with answers ranging from never to always.
  Raw scores are transformed to standardized T-score metrics, with a mean of 50 and standard deviation of 10
PROMIS Depression scale from baseline to study completion | 3 years
  Comparison of the PROMIS Depression scale at the end of follow-up to baseline. PROMIS tools were developed to be disease non-specific measures of health-related domains such as self-efficacy for symptom and medication management, depression, anxiety, fatigue, pain interference, sleep disturbance, and physical functioning. Each domain in composed of an item bank specific to a trait being measured. Item banks are calibrated on a common scale to facilitate comparability across varying populations. Depression is measured by various questions with answers ranging from never to always.
Comparison of Hospitlizations due to infections in the matched control and study group | 3 years
  Rate of hospitalizations, subcategorized for hospitalizations due to infections, compared between study participants and a matched control group
Comparison of rejection of matched control and study group | 3 years
  Incidence of treated rejections, compared between study participants and a matched control group
MRSB | 3 years
  Medication-Related Symptom Burden (MRSB), as defined as the change in number and severity of adverse effects
Graft survival at 3 years comparison of matched control vs. study group | 3 years
  Proportion of subjects with overall graft survival (including death with a functioning allograft) at year 3 post-transplant, compared between study participants and a matched control group
Graft survival at 1-2 years comparison of matched control vs. study group | 2 years
  Proportion of subjects with overall graft survival at year 1 and year 2 post-enrollment, compared between study participants and a matched control group
Graft loss during study period | 3 years
  Number of participants with graft loss, defined as permanent return to dialysis, retransplantation or patient death at any time during the 3-year primary follow-up study period;
Graft survival during study period | 3 years
  Graft survival calculated from the date of kidney transplantation until date of graft loss
Death-censored graft loss | 3 years
  Number of participants with death-censored graft loss, defined as permanent return to dialysis or retransplantation at any time during the 3-year primary follow-up study period. Patients who die with a functioning graft will be right censored
Patient death during study period | 3 years
  Number of participants with patient death from any cause at any time during the 3-year primary follow-up study period
Provider changes during study period | 3 years
  Rate of change in provider satisfaction from baseline to the end of follow-up using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patty West-Thielke, PharmD, Study Director — Transplant Genomics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli M, Wiebe N, Knoll G, Bello A, Browne S, Jadhav D, Klarenbach S, Gill J. Systematic review: kidney transplantation compared with dialysis in clinically relevant outcomes. Am J Transplant. 2011 Oct;11(10):2093-109. doi: 10.1111/j.1600-6143.2011.03686.x. Epub 2011 Aug 30. PMID 21883901
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LY, Albertus P, Ayanian J, Balkrishnan R, Bragg-Gresham J, Cao J, Chen JL, Cope E, Dharmarajan S, Dietrich X, Eckard A, Eggers PW, Gaber C, Gillen D, Gipson D, Gu H, Hailpern SM, Hall YN, Han Y, He K, Hebert H, Helmuth M, Herman W, Heung M, Hutton D, Jacobsen SJ, Ji N, Jin Y, Kalantar-Zadeh K, Kapke A, Katz R, Kovesdy CP, Kurtz V, Lavalee D, Li Y, Lu Y, McCullough K, Molnar MZ, Montez-Rath M, Morgenstern H, Mu Q, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Pearson J, Pisoni R, Plattner B, Port FK, Potukuchi P, Rao P, Ratkowiak K, Ravel V, Ray D, Rhee CM, Schaubel DE, Selewski DT, Shaw S, Shi J, Shieu M, Sim JJ, Song P, Soohoo M, Steffick D, Streja E, Tamura MK, Tentori F, Tilea A, Tong L, Turf M, Wang D, Wang M, Woodside K, Wyncott A, Xin X, Zang W, Zepel L, Zhang S, Zho H, Hirth RA, Shahinian V. US Renal Data System 2016 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2017 Mar;69(3 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2016.12.004. No abstract available. PMID 28236831
- [Background] Hart A, Smith JM, Skeans MA, Gustafson SK, Stewart DE, Cherikh WS, Wainright JL, Boyle G, Snyder JJ, Kasiske BL, Israni AK. Kidney. Am J Transplant. 2016 Jan;16 Suppl 2(Suppl 2):11-46. doi: 10.1111/ajt.13666. PMID 26755262
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Background] Lentine KL, Smith JM, Hart A, Miller J, Skeans MA, Larkin L, Robinson A, Gauntt K, Israni AK, Hirose R, Snyder JJ. OPTN/SRTR 2020 Annual Data Report: Kidney. Am J Transplant. 2022 Mar;22 Suppl 2:21-136. doi: 10.1111/ajt.16982. PMID 35266618
- [Background] El-Zoghby ZM, Stegall MD, Lager DJ, Kremers WK, Amer H, Gloor JM, Cosio FG. Identifying specific causes of kidney allograft loss. Am J Transplant. 2009 Mar;9(3):527-35. doi: 10.1111/j.1600-6143.2008.02519.x. Epub 2008 Feb 3. PMID 19191769
- [Background] Arms MA, Fleming J, Sangani DB, Nadig SN, McGillicuddy JW, Taber DJ. Incidence and impact of adverse drug events contributing to hospital readmissions in kidney transplant recipients. Surgery. 2018 Feb;163(2):430-435. doi: 10.1016/j.surg.2017.09.027. Epub 2017 Nov 22. PMID 29174434
- [Background] Couzi L, Moulin B, Morin MP, Albano L, Godin M, Barrou B, Alamartine E, Morelon E, Girardot-Seguin S, Mendes L, Misdrahi D, Cassuto E, Merville P. Factors predictive of medication nonadherence after renal transplantation: a French observational study. Transplantation. 2013 Jan 27;95(2):326-32. doi: 10.1097/TP.0b013e318271d7c1. PMID 23149477
- [Background] Gonzales HM, Fleming JN, Gebregziabher M, Posadas-Salas MA, Su Z, McGillicuddy JW, Taber DJ. Pharmacist-Led Mobile Health Intervention and Transplant Medication Safety: A Randomized Controlled Clinical Trial. Clin J Am Soc Nephrol. 2021 May 8;16(5):776-784. doi: 10.2215/CJN.15911020. Epub 2021 Apr 30. PMID 33931415
- [Background] Park S, Guo K, Heilman RL, Poggio ED, Taber DJ, Marsh CL, Kurian SM, Kleiboeker S, Weems J, Holman J, Zhao L, Sinha R, Brietigam S, Rebello C, Abecassis MM, Friedewald JJ. Combining Blood Gene Expression and Cellfree DNA to Diagnose Subclinical Rejection in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2021 Oct;16(10):1539-1551. doi: 10.2215/CJN.05530421. PMID 34620649
- [Background] Kalantar-Zadeh K, Kam-Tao Li P, Tantisattamo E, Kumaraswami L, Liakopoulos V, Lui SF, Ulasi I, Andreoli S, Balducci A, Dupuis S, Harris T, Hradsky A, Knight R, Kumar S, Ng M, Poidevin A, Saadi G, Tong A; World Kidney Day Steering Committee. Living well with kidney disease by patient and care-partner empowerment: kidney health for everyone everywhere. Kidney Int. 2021 Feb;99(2):278-284. doi: 10.1016/j.kint.2020.11.004. PMID 33509344
- [Derived] Fleming JN, Cober T, Hickey J, Stach L, Kawano A, Szczepanik A, Watson A, Imamura Y, Weems J, West-Thielke P. Clinical Utility of the OmniGraf Biomarker Panel in the Care of Kidney Transplant Recipients (CLARITY): Protocol for a Prospective, Multisite Observational Study. JMIR Res Protoc. 2022 Dec 14;11(12):e41020. doi: 10.2196/41020. PMID 36515980